CLINICAL TRIAL: NCT01223001
Title: Prevention of Depression and Enhancement of Cognitive Recovery Following Traumatic Brain Injury With Duloxetine
Brief Title: Feasibility Study of Duloxetine in the Treatment of Depression in Patients With Traumatic Brain Injury
Acronym: Duloxetine
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Most potential subjects had already been prescribed Cymbalta.
Sponsor: Rehabilitation Hospital of Indiana (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RHI 05-096; F1J-US-X025 (Other: Eli Lilly and Co.)
Record Dates: First submitted 2010-10-15; First posted 2010-10-18 (Estimated); Results first posted 2014-12-17 (Estimated); Last update posted 2014-12-17 (Estimated); Status verified 2014-11

CONDITIONS: Traumatic Brain Injury; Depression
Keywords: Depression; Traumatic brain injury; Duloxetine; Cymbalta; impaired cognitive function
MeSH Terms: conditions — Brain Injuries, Traumatic; Depression | interventions — Duloxetine Hydrochloride; Sugars; Lactose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Duloxetine (Active Comparator): Duloxetine 30 mg. PO daily to 120mg. PO daily for nine months in patients who have suffered a traumatic brain injury at least six months previously.
  Interventions: Drug: Duloxetine
- Sugar pill (Placebo Comparator): Sugar pills 30 mg. PO daily to 120mg. PO daily for nine months in patients who have suffered a traumatic brain injury at least six months previously.
  Interventions: Drug: Sugar pill

INTERVENTIONS:
Drug: Duloxetine — Duloxetine 30 mg. PO daily to 120mg. PO daily for nine months in patients who have suffered a traumatic brain injury at least six months previously.
  Other Names: Cymbalta
  Arms: Duloxetine
Drug: Sugar pill — Sugar pills 30 mg. PO daily to 120mg. PO daily for nine months in patients who have suffered a traumatic brain injury at least six months previously.
  Other Names: Lactose
  Arms: Sugar pill

SUMMARY:
The primary objective of the study is to compare the efficacy of duloxetine 60 mg by mouth daily with placebo in the prevention of depression associated with mild/moderate traumatic brain injury and to enhance cognitive function.

DETAILED DESCRIPTION:
The primary objective of the study is to compare the efficacy of duloxetine 60 mg by mouth daily with placebo in the prevention of depression associated with mild/moderate traumatic brain injury and to enhance cognitive function. Research exploring the use of selective serotonin reuptake inhibitors in the treatment of post-traumatic depression generally validates this approach (Horsfield et al., 2002). However, the literature suggests that serotonin/norepinephrine reuptake inhibitors such as duloxetine may be more effective in the treatment of depression.

ELIGIBILITY:
Inclusion Criteria:

* Study participants will be 40 men and women between the ages of 18 and 75 who provide appropriate consent and who are agreeable to study requirements
* Diagnosed with mild to moderate traumatic brain injury as defined by an initial Mayo Traumatic Brain Injury Severity Scale
* Have memory impairments defined by a Hopkins Verbal Learning Test delayed recall score which falls less than or equal to 1.5 standard deviation below the mean.

Exclusion Criteria:

* Refusal to give informed consent
* A previous Central Nervous System illness or injury, including seizure that exhibits residual symptoms.
* Current post-traumatic seizure disorder
* A previous diagnosis of a psychotic disorder
* Current or previous (in the last 6 months) treatment history for alcohol or substance dependency
* Medications affecting noradrenergic or dopaminergic systems, alpha-adrenergic antihypertensives, antidepressant, phenobarbital, Monoamine oxidase inhibitor (MAOI), scheduled benzodiazepines, psychoactive herbal supplements (including Kava, St. John's wort), or nutritional supplements or within at least 14 days of discontinuing treatment with the above medications or supplements.
* A known suicide risk
* A pregnant or breastfeeding woman
* Uncontrolled narrow-angle glaucoma
* Serious and/or unstable medical comorbidity (e.g., AIDS, cancer, history of uncontrolled hypertension or cardiovascular disease) psychological condition, or clinically significant laboratory abnormality that in the opinion of the investigator would compromise participation in the study or be likely to lead to hospitalization during the course of the study
* Liver enzymes > 1.5 times upper limit of normal
* Patients with end-stage renal disease (requiring dialysis) or severe renal impairment
* Known hypersensitivity to duloxetine or any of the inactive ingredients

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 1996-09; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lance Trexler, Ph.D., Principal Investigator — Rehabilitation Hospital of Indiana
Locations (1):
- Rehabilitation Hospital of Indiana, Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects recruited from in-patient and medical clinic population. All subjects suffering from traumatic brain injury and loss of cognitive function.
Pre-assignment Details: All subjects performed cognitive testing and assessment for depression. No subjects with seizure disorder or substance abuse issues or previous psychiatric history enrolled. Subjects excluded from the study had previously been prescribed Duloxetine.
Period: Overall Study
Arm/Group | Duloxetine | Sugar Pill
Started | 4 | 4
Completed | 0 | 0
Not Completed | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Duloxetine | Sugar Pill | Total
Number analyzed (Participants) | 4 | 4 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 4 | 8
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 4 | 3 | 7
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Hamilton Rating Scale for Depression
Description: To compare the efficacy of duloxetine 30 mg. PO daily to 120mg. PO daily with placebo in the prevention of depression associated with mild/moderate traumatic brain injury, utilizing the Hamilton Rating Scale for Depression (Hamilton, 1960; HAM-D) as the primary efficacy measure.
Time Frame: 9 months
Population: Analysis was not conducted. Study was terminated before interim analysis. Raw data is stored in a secure location, but not able to be accessed.
Arm/Group | Duloxetine | Sugar Pill
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Hopkins Verbal Learning Test
Description: To compare the effect of duloxetine vs. placebo on the recovery of memory functions of patients with traumatic brain injury, utilizing the 20-minute delayed recall score of the Hopkins Verbal Learning Test (Brandt, 1991) as the secondary efficacy measure.
Time Frame: 9 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Duration of study participation per subject.
Description: Subjects did not experience adverse events of any type.
Arm/Group | Duloxetine | Sugar Pill
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 0/4 | 0/4

LIMITATIONS AND CAVEATS:
All subjects excluded (n=6) had already been prescribed Duloxetine. Completion of the study by the remaining 4 per group was not achieved due to noncompliance.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days